CLINICAL TRIAL: NCT02297633
Title: System Evaluation of Reactive Oxygen Metabolites in the Value of Chronic Obstructive Pulmonary Disease
Brief Title: Evaluation of Reactive Oxygen Metabolites in the Value of COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Jie liu, Resident, Beijing Chao Yang Hospital
Other Study IDs: BJCYYT-12345
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: COPD(Chronic Obstructive Pulmonary Disease)
Keywords: COPD; reactive oxygen metabolites
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Stability in patients with COPD: Those patients diagnosed COPD according to the GOLD guideline and without acute exacerbation within one month.
- AECOPD: the diagnosis of an exacerbation relies exclusively on the clinical presentation of the patient complaining of an acute change of symptoms (baseline dyspnea, cough, and/or sputum production) that is beyond normal day-to-day variation.
- Healthy persons without smoking: The healthy people who do not smoke
- Healthy persons with smoking: Healthy persons who smoke

SUMMARY:
This study through the long-term observation followed up for 2 years to find the change of the COPD patients blood ROMs, systematically evaluate the relationship between ROMs and the severity of COPD. Evaluate the differences of prognosis between the different oxidative stress level (according to the level of ROMs are divided into higher and normal phenotype). Explore the new oxidative stress evaluation index ROMs application value in COPD.

DETAILED DESCRIPTION:
Reactive oxygen metabolites (reactive oxygen metabolites, ROMs) test is a method by measuring the total reactive oxygen metabolites (ROMs) content in blood so as to evaluate the overall level of oxidative stress in the human body .Our previous studies have established the method of detecting ROMs which is suitable for fully automatic biochemical analyser.Our study through the long-term observation followed up for 2 years to find the change of the COPD patients blood ROMs, systematically evaluate the relationship between ROMs and the severity of COPD. Evaluate the differences of prognosis between the different oxidative stress level (according to the level of ROMs are divided into higher and normal phenotype). Explore the new oxidative stress evaluation index ROMs application value in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD according to GOLD 2013

Exclusion Criteria:

* A history of asthma or other chronic lung diseases Take Antioxidant therapy There are new or recurrent symptomatic myocardial ischemia, severe arrhythmia, cardiac insufficiency cerebrovascular disease Senile dementia or cognitive impairment cancer Severe liver and kidney and other viscera function insufficiency Language communication barriers Limb activity disorder The last 3 months participated in sports training

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chaoyang hospital clinic
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The different levels of the ROMs among different groups | 3 years
  Apply the analysis of variance to compare the different levels of ROMs among the four different groups

SECONDARY OUTCOMES:
The differences of the ROMs among the different lung function levels in the stable stage of COPD group | 3 years
  Apply the analysis of variance to compare the differences of the ROMs among the lung function levels in the stable stage of COPD group.
The relevance of the ROMs with the lung function levels in the stable stage of COPD group | 3 years
  Apply Pearson correlation to compare relevance the of the ROMs with the lung function levels in the stable stage of COPD group.
The relevance of the ROMs with the score of mMRC in the stable stage of COPD group | 3 years
  Apply Pearson correlation to compare relevance the of the ROMs with score of mMRC in the stable stage of COPD group.
The relevance of the ROMs with the score of CAT in the stable stage of COPD group | 3 years
  Apply Pearson correlation to compare relevance the of the ROMs with score of CAT in the stable stage of COPD group.
The relevance of the ROMs with the numbers of exacerbation in the stable stage of COPD group | 3 years
  Apply Pearson correlation to compare relevance the of the ROMs with numbers of exacerbation in the stable stage of COPD group.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Yang, Doctor, Study Director — Respiratory Institute, Beijing chaoyang hospital
Locations (1):
- Respiratory Institute;Beijing chaoyang hospital, Beijing, Beijing Municipality, China